CLINICAL TRIAL: NCT03992794
Title: ADAPTED: Assessment of Disease Severity, Progression and Treatment in Infected Patients Presenting to the Emergency Department
Brief Title: Assessment of Disease Severity, Progression and Treatment in Infected Patients Presenting to the Emergency Department
Acronym: ADAPTED
Status: Completed | Type: Observational
Sponsor: Juan González-del Castillo (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor-Investigator, Juan González-del Castillo, HEAD OF INFECTION DISEASE GROUP OF SPANISH EMERGENCY MEDICINE SOCIETY, Sociedad Española de Medicica de Emergencias
Organization: Sociedad Española de Medicica de Emergencias (Other)
Other Study IDs: 18/081-E
Record Dates: First submitted 2019-06-16; First posted 2019-06-20 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Sepsis
Keywords: Sepsis; Emergency department; Sepsis biomarkers; MR-proADM
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total patients: Consecutive patients presenting to the ED with either a suspected or documented infection in which blood samples were taken during routine. An extra blood sample was taken to measure PCT & MR-proADM using the Samsung IB10 point of care assay.
  Interventions: Diagnostic Test: Measurement of MR-proADM

INTERVENTIONS:
Diagnostic Test: Measurement of MR-proADM — It is an observational study. The only intervention was the measure of MR-proADM, but no clinical decision was made based on its value, since the physician attending the patient did´n know the value of MR-proADM

SUMMARY:
The results of the SIDED study (doi: 10.1186 / s13054-019-2329-5) showed that MR-proADM can be a good biomarker to establish the prognosis of patients attended in the emergency department (ED) due to suspected infection. MR-proADM could be useful to help making-decision regarding admission or discharge of patients, and in addicion to determine the need to apply or not early antibiotic treatment. However, despite analyzing more than 2,500 patients from 8 countries, the original study had a number of limitations. Samples of the biomarkers were retrospectively analyzed in a device that is not routinely used in the ED (Kryptor, Thermo Fisher, Germany). The availability of MR-proADM at the point of care could facilitate its widespread use in all EDs. This study is conducted to confirm the results of the SIDED study by using a device at the patient's bedside that allows the quantitative determination of the MR-proADM and procalcitonin biomarkers, instead of using a Kryptor platform.

DETAILED DESCRIPTION:
Despite significant improvements in diagnostic and preventative measures, the incidence of sepsis has continued to escalate rapidly in hospitalized patients, with mortality rates ranging between 10 - 54%, depending on the level of severity. The earliest possible identification and assessment of sepsis patients entering the Emergency Department (ED) is therefore crucial in providing the patient with the most appropriate management and treatment strategy at the earliest time point possible. Indeed, an early identification of patients with an infection and at a high risk of cardiovascular and organ dysfunction can lead to an earlier individualised treatment, a potential reduction in the number of clinical complications, and an overall decrease in hospital mortality.

Adrenomedullin (ADM), a 52 amino acid peptide, is a member of the calcitonin peptide family and is widely expressed in many tissues and organs, although its main sources of production include the endothelial and vascular smooth muscle cells. Adrenomedullin can act as both a hormone and cytokine (often termed a "hormokine") in an autocrine and paracrine manner, and its potent vasodilatory and hypotensive response is elicited through an initial increase in cyclic adenosine monophosphate levels, and a subsequent production of nitric oxide.

The importance of adrenomedullin in homeostasis is illustrated by its central role in the up- and down-regulation of cytokines and other mediators, as well as its own stimulatory and inhibitory effect on cytokine production. Indeed, Interleukin (IL)-1β and tumour necrosis factor (TNF) are two of the most potent stimulators for adrenomedullin production and adrenomedullin itself is up-regulated by hypoxia, bacterial products and shear stress, amongst many other factors.

Finally, adrenomedullin has been shown to have a variety of physiological functions, including immune-modulating, direct bactericidal, diuretic and potent vasodilatory activity, and in healthy conditions, circulates at low picomolar concentrations. However, plasma levels are significantly up-regulated in many diseased states in proportion to disease severity such as hypertension, renal failure, lower respiratory diseases and septic shock, due to either damage to the endothelial cells or microvascular and microcirculatory impairment.

This allows clinicians to determine the patients most at risk of developing complications upon their admission to the ED or ICU, in order to rapidly triage and administer the most effective treatment, in the shortest space of time.

However, reliable measurement of ADM is challenging due to a number of issues, such as a short half life of 22 minutes, rapid degradation by proteases and binding to complement factor H. The measurement of its stable precursor molecule, MR-proADM, provides a solution to these problems, since reliable measurements in relation to adrenomedullin can be made in a 1:1 ratio, thus allowing changes in protein concentrations to be determined.

The majority of deaths in patients suffering from sepsis occur due to multiple organ failure, related to the primary infection. However, complications leading up to initial organ dysfunction and failure include factors such as an impaired microcirculation, enhanced microvascular permeability, a decrease in the number of perfused capillaries, endothelial cell apoptosis and an abnormal systemic blood flow to organ systems. Few tools currently available have the ability to accurately assess these early physiological changes.

The vasodilatory and microcirculatory properties of adrenomedullin are therefore of significant importance during the pathophysiology and progression of sepsis, with increased levels being shown to lead to a decreased vascular resistance and a significantly increased microvascular blood flow in the liver, small intestine, kidney and spleen. Indeed, the production of adrenomedullin has been shown to have:

* protective properties against endothelial permeability and consequent organ damage
* protective effects in organs in response to bacterial induced shock
* the ability to stabilize the microcirculation in inflammation - a hallmark of organ failure
* the ability to restore endothelial stability in infected organs due to prevention of undesired inflammatory decompartmentalization.

Crucially, the body can facilitate the localized cellular production and release of adrenomedullin in order to meet the specific perfusion requirements of individual organs, which can be crucial in maintaining blood supply.

Whilst current benchmarks of sepsis which include lactate and SOFA scores can accurately assess the degree of tissue hypoxia and organ dysfunction at any given time point, elevated MR-proADM levels can accurately reflect the early microvascular changes that occur in the build up to subsequent organ damage and dysfunction, the majority of which are extremely difficult to detect using standard clinical techniques, biomarkers or severity scores.

The clinical use of MR-proADM

Thus, MR-proADM levels can provide the treating physician with an accurate reflection of abnormalities in the microcirculation before the patient develops any form of organ dysfunction or adverse clinical signs become apparent, thus providing an earlier warning of any developing complications associated with the infectious condition. Indeed, even when diagnostic biomarkers such as PCT, CRP or lactate are either initially low or decreasing satisfactorily, patients might still be at considerable risk of further complications, which can be highlighted through elevated MR-proADM values. In these cases, an immediate transfer to a more intensive ward or department and an early, rapid and goal directed therapeutic treatment would most likely be required in order to achieve the best possible clinical outcome for the patient.

On the other hand, resolving issues in the microcirculation/endothelium can be indicative of an improvement in clinical status, and illustrated by low MR-proADM values. Accordingly, even in the presence of elevated laboratory or other biomarker values and poor clinical signs, the patient in question may develop no further physiological complications apart from the pre-existing microbial infection itself, which when treatment is correctly initiated, can facilitate an earlier transfer onto a less acute ward, consequently saving the healthcare provider valuable resources such as physician time, hospital beds and overall financial budget.

The results of the SIDED study (doi: 10.1186 / s13054-019-2329-5) showed that MR-proADM measurement at presentation could accurately assess disease severity and identify specific patient populations based on the likelihood of subsequent disease progression. This was of particular importance in patients with few pathophysiological signs and symptoms, as indicated by low SOFA, qSOFA or NEWS scores, where initial treatment may either be withheld, delayed or insufficient. Our study therefore, for the first time, highlights the use of MR-proADM in potentially identifying this patient population in order to initiate appropriate treatment strategies at the earliest opportunity.

Based on the results of this study, two clinically important uses for MR-proADM can be proposed: (i) an early escalation of treatment in patients with MR-proADM concentrations ≥1.5 nmol/L, thus identifying an already high level of disease severity or a high potential for further development and progression, and (ii) a decreased number of hospital admissions allowing a safe increase in out-patient treatment in patients with MR-proADM concentrations <0.9 nmol/L.

Samples of the biomarkers were in SIDED study retrospectively analyzed in a device that is not routinely used in the ED (Kryptor, Thermo Fisher, Germany). The availability of MR-proADM at the point of care could facilitate its widespread use in all EDs. This study is conducted to confirm the results of the SIDED study by using a device at the patient's bedside (Samsung IB10 platforms) that allows the quantitative determination of the MR-proADM and procalcitonin biomarkers, instead of using a Kryptor platform, and obtaining the biomarkers results in no more than 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Consecutive patients presenting to the ED with either a suspected or documented infection
* Blood samples taken during routine use only
* Patient has given written informed consent

Exclusion Criteria:

* Age < 18 years
* Patients where no blood samples were taken for routine purposes
* Those with no suspicion of infection
* Pregnancy
* Refusal to participate
* Patient has already participated in a similar clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED with either a suspected or documented infection
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Mortality
ICU admission | 28 days
  Intensive care admission of the attended patient
Time of antibiotic administration | 24 hrs
  Length of time from initial presentation at the ED to the first dose of antibiotics being administered.

SECONDARY OUTCOMES:
Disease progression | 28 days
  Composite endpoint consisting of infection-related 30-day mortality, ICU admission and a ≥2 point increase in NEWS or SOFA score between presentation and 72 hrs
Hospital readmission | 28 days
  Hospital readmission

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gonzalez del Castillo, MD, phD, Principal Investigator — Head of Infection Disease Group of Spanish Emergency Medicine Society
Locations (3):
- Spain (3):
  - Hospital Universitario General de Alicante, Alicante
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospita Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saeed K, Wilson DC, Bloos F, Schuetz P, van der Does Y, Melander O, Hausfater P, Legramante JM, Claessens YE, Amin D, Rosenqvist M, White G, Mueller B, Limper M, Callejo CC, Brandi A, Macchi MA, Cortes N, Kutz A, Patka P, Yanez MC, Bernardini S, Beau N, Dryden M, van Gorp ECM, Minieri M, Chan L, Rood PPM, Del Castillo JG. The early identification of disease progression in patients with suspected infection presenting to the emergency department: a multi-centre derivation and validation study. Crit Care. 2019 Feb 8;23(1):40. doi: 10.1186/s13054-019-2329-5. PMID 30736862